CLINICAL TRIAL: NCT04108286
Title: Ex-vivo Adhesion of Bacteria to Different Contact Lens Materials
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn due to COVID-19 and country restrictions
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-6333
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects that are habitual wearers of spherical soft contact lenses will be randomly assigned to 1 of 2 contralateral lens sequences (Right: TEST/ Left: CONTROL) or (Right: CONTROL/ Left: TEST).
  Interventions: Device: 1-DAY ACUVUE MOIST; Device: DAILIES AQUA COMFORT PLUS
- CONTROL/TEST (Experimental): Eligible subjects that are habitual wearers of spherical soft contact lenses will be randomly assigned to 1 of 2 contralateral lens sequences (Right: TEST/ Left: CONTROL) or (Right: CONTROL/ Left: TEST).
  Interventions: Device: 1-DAY ACUVUE MOIST; Device: DAILIES AQUA COMFORT PLUS

INTERVENTIONS:
Device: 1-DAY ACUVUE MOIST — TEST
  Other Names: 1DAM
Device: DAILIES AQUA COMFORT PLUS — CONTROL
  Other Names: DACP

SUMMARY:
This is a single-site, 4-visit, contralateral, dispensing, open-label, randomized study. Each eligible subject will be randomized into one of two sequence groups to wear two lens types contralaterally (Test on the right eye and Control on left eye or vice versa).

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study.

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 45 (inclusive) years of age at the time of screening.
  4. Be a current spherical soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.
  5. Have a pair of spectacles with corrected vision of 20/40 or better in each eye or uncorrected vision is 20/40 or better in each eye
  6. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 through -6.00 D in each eye.
  7. The subject has a best-corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study.

  1. Currently pregnant or breastfeeding.
  2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
  3. Any autoimmune disease or use of medication, which may interfere with contact lens wear. Habitual medications used by successful soft contact lens wearers are considered acceptable.
  4. Any ocular abnormalities such as entropion, ectropion, extrusions, chalazia, recurrent styes, history of recurrent corneal erosions.
  5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  6. Multifocal, toric or extended wear contact lens correction.
  7. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  8. History of binocular vision abnormality or strabismus.
  9. Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report.
  10. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  11. Any ocular infection.
  12. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the EFRON scale (Appendix G), any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
  13. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-01-06 (Estimated); Study Completion 2021-01-06 (Estimated)

PRIMARY OUTCOMES:
Bacterial adhesion of clinical isolates of P. aeruginosa | up to 2-week follow-up
  Evaluation of the bacterial adhesion of 2 strains of bacteria, P. aeruginosa, on worn lenses based on the number of viable bacteria on the lens measured in colony forming unit (CFU).

SECONDARY OUTCOMES:
Uptake of Lysozyme on worn lenses | up to 2-week follow-up
  Uptake of Lysozyme on worn lenses: Evaluation of the uptake of lysozyme between different lens materials of worn lenses based on the clearance zone measured in the nearest (mm).

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu